CLINICAL TRIAL: NCT03743883
Title: Effectiveness of Low-dose Aspirin in Gastrointestinal Cancer Prevention -United Kingdom ("ENgAGE - UK"): A Cohort Study on the Risk of Gastric and Oesophageal Cancer Among New Users of Low-dose Aspirin Using the THIN Database in the UK
Brief Title: EffectiveNess of Low-dose Aspirin in Prevention of Cancer in the Stomach and Oesophagus (GastrointEstinal Cancer Prevention) - United Kingdom ("ENgAGE - UK"): Study to Evaluate the Risk of Cancer in the Stomach and Oesophagus Among New Users of Low-dose Aspirin Using the THIN Database in the UK
Acronym: ENgAGE-UK
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20326
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Prevention of Oesophagus Cancer and Stomach Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low-dose ASA cohort: A person is identified as newly exposed to low-dose ASA, he/she will become member of new user low-dose ASA cohort and that date will be the start date for outcome follow-up.
  Interventions: Drug: Acetylsalicylic Acid(BAYE4465, Aspirin )
- Comparison unexposed cohort: When a member of new user low-dose ASA cohort is confirmed, one comparison member will be confirmed also from the source population not yet censored on that day (start date) and with the same distribution of matching factors (age, sex, time interval since entry date and number of PCP visits in the year prior to start date) of its low-dose ASA pair with the only difference of being free of ASA on start date.

INTERVENTIONS:
Drug: Acetylsalicylic Acid(BAYE4465, Aspirin ) — Administration according to clinical practice
  Groups: Low-dose ASA cohort

SUMMARY:
Researchers already did studies in low-dose Aspirin for the prevention of heart and blood vessels disease and for the prevention of cancer of the colorectum. In this study, they want to learn whether an effect for the prevention of oesophagus cancer and stomach cancer goes along with the use of low-dose ASA on patients taking this medicine for the prevention of heart and blood vessels disease compared to non-use. To find this out electronic medical records stored in primary care database in the UK, The Health Improvement Network (THIN), will be used.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-89 years
* Enrolled with the PCP for at least 2 years
* To have a history of computerized prescriptions in THIN for at least 1 year prior to start date

Exclusion Criteria:

* To be exposed to low-dose ASA before entering in the study
* Having a diagnosis of any cancer before entering in the study

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population will be constituted (inclusion criteria) by individuals who are aged 40-89 years in the THIN database in the UK, who are enrolled with the primary care doctor (PCP) for at least 2 years, or have a history of computerized prescriptions for at least 1 year prior to start date and who are free of low-dose ASA and cancer to become a member of the source population.
Sampling Method: Non-Probability Sample
Enrollment: 99999 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence rates of oesophageal cancer and stomach cancer with use of low-dose ASA overall compared to non-use | Retrospective analysis between 1-Jan-2005 and 31-Dec-2017
  Diagnosis of cancer is routinely recorded by means of Read codes in THIN database
Incidence rates of oesophageal cancer and stomach cancer with use of low-dose ASA by age compared to non-use | Retrospective analysis between 1-Jan-2005 and 31-Dec-2017
  Age: 40-64 years, 65-74 years and 75 and more years.
Incidence rates of oesophageal cancer and stomach cancer with use of low-dose ASA by sex-specific compared to non-use | Retrospective analysis between 1-Jan-2005 and 31-Dec-2017
  Sex: Male, Female

SECONDARY OUTCOMES:
Incidence of oesophageal cancer and stomach cancer among new users of low-dose ASA | Retrospective analysis between 1-Jan-2005 and 31-Dec-2017
Duration of low-dose ASA | Retrospective analysis between 1-Jan-2005 and 31-Dec-2017
  Duration of treatment will be calculated among current users.
Dose-response of low-dose ASA | Retrospective analysis between 1-Jan-2005 and 31-Dec-2017
  The following daily doses will be ascertained: 75 mg, 150 mg and 300 mg.
Number of case-fatality of oesophageal cancer and stomach cancer among new users of low-dose ASA | Retrospective analysis between 1-Jan-2005 and 31-Dec-2017
Incidence of oesophageal cancer and stomach cancer among new users of low-dose ASA for primary or secondary cardiovascular prevention | Retrospective analysis between 1-Jan-2005 and 31-Dec-2017
  The primary and secondary cardiovascular prevention population of low-dose ASA users will be defined using a computer algorithm ascertaining any recorded Read code suggestive of cardiovascular disease (CVD).

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com